CLINICAL TRIAL: NCT07402265
Title: Piloting a Brief, Online Intervention for Suicidality in Sexual and Gender Minority Youth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University (Other)
Collaborators: Western University, Canada (Other); Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Lindsay P. Bodell, PhD, Associate Professor, Western University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 127209
Record Dates: First submitted 2026-01-30; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Suicidal Thoughts; Sexual and Gender Minorities; Youth
Keywords: Suicidal thoughts; Sexual and Gender Minorities; Youth; Brief; Online; Self-Guided; Self-Compassion; Self-Neutrality
MeSH Terms: conditions — Suicidal Ideation; Coitus

STUDY DESIGN:
Intervention Model Description: All participants will complete the same program. There is no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will complete the online, self-guided program, which will take approximately 30 minutes and involve participants completing modules describing how to use self-compassion/self-neutrality techniques to reduce suicidal thoughts.
  Interventions: Behavioral: KindMind

INTERVENTIONS:
Behavioral: KindMind — This intervention is hosted on Wix-com and involves multiple self-guided modules in which participants are taught how to use self-compassion and/or self-neutrality to reduce suicidal thoughts. This intervention is tailored to sexual and gender minority youth.

SUMMARY:
Sexual and gender minority youth (i.e., LGBTQ+ individuals) are at elevated risk for suicidal thoughts compared to cisgender/heterosexual youth and there is increased demand for programs and treatments tailored to this population. The current study seeks to pilot a brief, online, self-guided intervention for suicidal thoughts designed for sexual and gender minority youth to test if this intervention is acceptable to this population and if completing this intervention significantly decreases suicidal thoughts.

DETAILED DESCRIPTION:
The current study will pilot an intervention for suicidal thoughts in sexual and gender minority youth. We will recruit of a sample of sexual and gender minority youth who report experiencing recent thoughts of suicide. Participants will be asked to complete a battery of questionnaires including demographic questions and mental health symptom assessments, then complete the intervention, and finally complete additional questionnaires. One month after completing the intervention, participants will be asked to complete a series of questionnaires. This study is designed to evaluate the acceptability and initial effectiveness of this intervention and will not include a control group.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Canada
* Fluent in English
* Youth (i.e., 13-25 years)
* Identifies as a sexual and/or gender minority (i.e., any sexual identity excluding heterosexual and/or any gender identity excluding cisgender)
* Endorses experiencing any suicidal ideation within the past 6 months
* Access to a computer and able to participate virtually

Exclusion Criteria:

* Does not meet the inclusion criteria

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants must identify as a sexual and/or gender minority to participate. All genders are eligible if the individual meets the other inclusion criteria (e.g., identifies as either a sexual minority or gender minority).
Enrollment: 250 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation Questionnaire - Junior | From Baseline (i.e., before intervention administration) to four weeks after intervention administration.
  Suicidal Ideation Questionnaire - Junior (SIQ-Jr; Reynolds, 1987). The SIQ-Jr was used to assess suicidal ideation in the current study. This self-report measure include 15 items of suicidal thoughts that are rated on a 7-item scale (i.e., Almost every day, couple of times a week, about once a week, couple of times a month, About once a month, I had this thought before but not in the past month, I never had this thought) of how frequency the respondent had each thought in their mind over the past month. Sample items include I thought about dying, I wished I were dead, and I thought about killing myself. The SIQ-Jr is scored by summing the responses to create a total score from 0-90, with higher scores indicating a higher severity of suicidal ideation.

SECONDARY OUTCOMES:
Suicidal Ideation Thoughts and Behaviours Interview - Revised | From Baseline (i.e., before intervention administration) to four weeks after intervention administration.
  Suicidal Ideation Thoughts and Behaviours Interview - Revised (SITBI -R; Gratch et al., 2022). Select items from the SITBI-R will be administered to capture suicidal behaviour, including frequency and severity of suicide attempts.
Self-Compassion Scale - Short Form | From Baseline (i.e., before intervention administration) to four weeks after intervention administration.
  Self-Compassion Scale - Short Form (SCS-SF; Raes et al., 2011). The SCS-SF is a 12-item measure that assesses trait self-compassion. Each item is rated on a 5-point scale of how the participant typically reacts to themselves during difficult times, ranging from Almost never to Almost Always. Six subscales are computed corresponding to the six components of self-compassion based on Neff's (2003) conceptualization: Self-Kindness, Self-Judgement, Common Humanity, Isolation, Mindfulness, and Overidentification. A total score is computed by averaging the six subscale total scores. Higher scores indicated higher self-compassion. Sample items include I try to see my failing as part of the human condition and I'm disapproving and judgmental about my own flaws and inadequacies.
Patient Health Questionnaire - 9 | From Baseline (i.e., before intervention administration) to four weeks after intervention administration.
  Patient Health Questionnaire - 9 (PHQ-9; Kroenke et al., 2001). The PHQ-9 a self-report assessment of depressive symptoms. The PHQ-9 includes nine items that ask participants to rate how frequently they experienced each problem (i.e., Little interest or pleasure in doing things, Feeling tired or having low energy) over the past two weeks, with a 4-point scale of frequency (i.e., Not at all, Several days, More than half the days, Nearly every day). A total score is summed and can range from 0-27. Higher total scores indicate greater severity of depressive symptoms. An additional item not included in the total score asks participants to rate how difficult the problems they indicated make it for them to do work, take care of things at home, and get along with other people.
Hopelessness Scale for Children | From Baseline (i.e., before intervention administration) to four weeks after intervention administration.
  Hopelessness Scale for Children (HSC; Kazdin et al., 1983). The HSC includes 17 true/false items assessing hopelessness in children as young as 5 years old. Total scores are summed and the higher the total score, the greater the hopelessness for the future. Sample items include I will have more good times than bad times and I don't think I will get what I really want.
Generalized Anxiety Disorder - 7 | From Baseline (i.e., before intervention administration) to four weeks after intervention administration.
  Generalized Anxiety Disorder - 7 (GAD-7; Spitzer et al., 2006) . The GAD-7 is a self-report assessment of anxiety. The respondent indicates how often they have experienced each of seven listed symptoms over the past two weeks, including items such as Not being able to stop or control worrying and Becoming easily annoyed or irritable. Items are rated on a 4-point scale of frequency (i.e., Not at all, Several days, More than half the days, Nearly every day). Total scores range from 0-21, with higher scores indicating higher severity of anxiety. An additional item not included in the total score asks participants to rate how difficult the problems they indicated make it for them to do work, take care of things at home, and get along with other people.
Difficulties in Emotion Regulation Scale - Short Form | From Baseline (i.e., before intervention administration) to four weeks after intervention administration.
  Difficulties in Emotion Regulation Scale - Short Form (DERS-SF; Kaufman et al., 2016). The DERS-SF is a self-report measure of difficulties regulating emotion. This measure has 18 items that are rated on a 5-point scale assessing how often each item applies to the participant, including the following options: Almost never (0-10%), Sometimes (11-35%), About half of the time (36-65%, Most of the time (66-90%), and Almost always (91-100%). The DERS-SF includes items such as When I'm upset, I have difficulty concentrating and I pay attention to how I feel. A total score and six subscale scores (Strategies, Nonacceptance, Impulse, Goals, Awareness, Clarity) are created by adding item scores and higher scores reflect greater difficulties with emotion regulation. Total scores range from 18-90.

OTHER OUTCOMES:
Intervention Feedback Questions. | Immediately following intervention administration
  After the intervention, participants will be asked several unstandardized feedback questions rated on a 5-point Likert Scale (i.e., Strongly Disagree, Disagree, Neither Agree or Disagree, Agree, Strongly Agree) about how acceptable, helpful, and engaging the intervention is. Participants will also be asked how likely to use the intervention they would be and how likely they are to recommend it to a friend.
Visual Analogue Scales | From immediately before intervention administration to immediately after intervention administration.
  Visual Analogue Scales (VAS). VAS are a measurement method that involves participants marking a point on a continuous line between two extreme points to indicate the intensity of a feeling or mood. For this study, all VAS involved a slider scale in which the participant could indicate a value between 0 and 100, with lower scores indicating lower intensity and higher scores indicating higher intensity. For example, to measure state sadness, participants were given the following instructions: Using the slider below, please indicate how sad you feel in this moment. Scores can range from 0-100. Lower scores indicate less sadness and higher scores indicate more sadness. VAS will be used to assess state self-compassion, self-neutrality, hopelessness, distress, anger, anxiety, sadness, tiredness, and desire to self-harm immediately before and after completing the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay P Bodell, PhD, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified IPD that is included in the published results of the study will be shared.